CLINICAL TRIAL: NCT03709017
Title: Post-Marketing Surveillance of Safety and Effectiveness of Iclusig® Tablets in Korean Patients With CML or Ph+ ALL Under the "Risk Management Plan"
Brief Title: Iclusig PMS in CML or Ph+ALL Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 297-402-00002
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ponatinib — Iclusig 45mg, 15mg
  Other Names: Iclusig

SUMMARY:
This is a Post-Marketing Surveillance (PMS) of Iclusig® Tablets in accordance with Korean regulations on Risk Management Plan (RMP). This PMS is to assess safety and effectiveness data after administrating Ponatinib (of Iclusig® Tablets) per approved indication, usage and dosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed Iclusig® per Prescribing information (PI) for the purpose of treatment

Exclusion Criteria:

* Patients with known or suspected hypersensitivity to ponatinib or to any ingredient of the drug
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed Iclusig® tablets and provide written informed consent will be enrolled. The number of patients to be enrolled by each investigator will vary.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The incidence rate and the number of Adverse Events (AE)/Adverse Drug Reactions (ADR), Serious AE/ADR, Unexpected AE/ADR | until 14 days after last administration

SECONDARY OUTCOMES:
The number of subjects who satisfy CHR | at 3 months and 6 months from administration
The percentage of subjects who satisfy CHR | at 3 months and 6 months from administration
The number of subjects who satisfy MCyR | at 3 months and 6 months from administration
The percentage of subjects who satisfy MCyR | at 3 months and 6 months from administration
The number of subjects who satisfy MMR | at 3 months and 6 months from administration
The percentage of subjects who satisfy MMR | at 3 months and 6 months from administration

CONTACTS AND LOCATIONS:
Locations (1):
- Kosin University Gaspel Hospital, Busan, South Korea